CLINICAL TRIAL: NCT04603274
Title: Efficacy of Electroacupuncture in Carpal Tunnel Syndrome: a Clinical, Electrophysiologic and Ultrasonographic Study
Brief Title: Efficacy of Electroacupuncture in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aretaieion University Hospital (Other)
Collaborators: University of West Attica (Other); Lilian Voudouri Foundation (Unknown)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Professor of Anesthesiology, Aretaieion University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 233/30-06-2020 electroacup
Record Dates: First submitted 2020-10-18; First posted 2020-10-26 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Carpal Tunnel; Carpal Tunnel Syndrome; Pain; Pain Syndrome; Pain Syndrome Myofascial
MeSH Terms: conditions — Median Neuropathy; Carpal Tunnel Syndrome; Pain; Somatoform Disorders; Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- upper extremity diagnosed with carpal tunnel syndrome (Other): 8 sessions of electroacupuncture, 2 days a week for 1 month by experienced physicians
  Interventions: Procedure: 8 sessions of electroacupuncture to the upper limb with carpal tunnel syndrome

INTERVENTIONS:
Procedure: 8 sessions of electroacupuncture to the upper limb with carpal tunnel syndrome — All participants will accept 8 sessions of electroacupuncture, 2 days a week for 1 month by experienced physicians. Acupuncture sterile disposable needles 0,25x 0,25 mm will be inserted for 20 minutes at specific acupuncture points to all patients. Electrical stimulation will be applied at specific acupuncture points for 20 minutes.

SUMMARY:
The aim of this clinical study is to assess the effectiveness of electroacupuncture in reducing the severity of symptoms, in improving limb function, in improving the aesthetic and motor conduction of the median nerve and in reducing its cross-sectional area at the inlet of the carpal tunnel in patients with carpal tunnel syndrome. All upper extremities diagnosed with carpal tunnel syndrome will be treated with electroacupuncture for 8 sessions. Clinical, electrophysiological and ultrasonography outcome measures will be evaluated before and after the intervention, to assess the result.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common mononeuritis, with a significant burden on both patients and public health. For mild and moderate cases, conservative methods, including immobilization, corticosteroid injections, oral medications and physical therapy have been suggested as appropriate treatments, with mixed results. Acupuncture and related therapies has been used worldwide over the last few years in the management of CTS, with generally positive results. However, more studies will be needed to assess the role of acupuncture as an independent therapeutic modality to CTS.

This is a clinical study that will be conducted in the pain clinic at the department of Anaesthesiology of Aretaieion University Hospital as well as in the Laboratory of Musculoskeletal Physiotherapy of University of West Attica, with which there is a cooperation agreement. All recruited participants will be treated with the same acupuncture protocol at the limb that will be diagnosed with carpal tunnel syndrome. If the patients are diagnosed with bilateral CTS, both wrists will be treated. Clinical, electrophysiological and ultrasonography outcomes will be measured before and after the intervention.

In order to record the possible influence of psychosomatic characteristics, the Greek version of the Hospital Anxiety & Depression (HAD) Scale will be used before the treatment. As a result the anxiety and the depression of the participants will be quantified with a simple clinical tool.

All participants will accept 8 sessions of electroacupuncture, 2 days a week for 1 month by experienced physicians.

All participants in the study will be evaluated 3-7 days before and 3-7 days after the treatment protocol with clinical, electrophysiological and ultrasonographical outcome measures. In patients with bilateral symptoms, each limb will be assessed separately.

ELIGIBILITY:
Inclusion Criteria:

* paraesthesia, numbness, pain in the area of distribution of the median nerve
* worsening of symptoms at night or with repeated movements of the wrist
* aesthetic or/and motor deficits in the area of distribution of the median nerve
* Median sensory nerve conduction velocity (SNCV), first digit to wrist <42 m/s
* Median distal motor latency (DML), wrist to thenar eminence >4 ms.
* Difference between the median and radial sensory latencies to the thumb ≥ 0,5 ms.
* Median palmar peak latency (PL)> 2,2 ms and in comparison to ulnar palmar peak latency ≥ 0,4 ms.
* Median versus Ulnar - Lumbrical - Interossei studies (Difference between the median 2nd lumbrical & ulnar 1st palmar interosseous distal latency, >0,5 ms).

Exclusion Criteria:

* age<18 years
* absence of the above electrophysiological criteria
* diagnosis of another disease during the electrophysiological test
* patients with severe carpal tunnel syndrome to be operated on
* thenar muscle atrophy
* previous carpal tunnel release surgery
* local steroid injections in the last 3 months
* clinical active rheumatic disease
* diabetic polyneuropathy
* alcoholism
* neurological disease affecting the upper extremity (stroke, multiple sclerosis, amyotrophic lateral sclerosis, cervical radiculopathy, polyneuropathy)
* contraindications to electroacupuncture: pacemaker, epilepsy, skin disorders in the upper extremities
* no consent to the study
* language or communications barriers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
change from baseline in Symptom Severity Scale (SSS) of -the Greek- Boston carpal tunnel questionnaire (BCTQ) | 3-7 days after the treatment protocol
  The Boston carpal tunnel questionnaire (BCTQ) is an easy, disease-specific measurement of self-reported symptom severity and functional status for carpal tunnel syndrome (CTS). It has two distinct scales, the Symptom Severity Scale (SSS) which has 11 questions and the Functional Status Scale (FSS) containing 8 questions. Each scale using a five-point rating score generates a final score which ranges from 1 to 5, with the higher indicating greater disability. We will use the Greek version of the BCTQ, which had been examined for reliability and validity and responsiveness before and after the intervention.

SECONDARY OUTCOMES:
change from baseline in Functional Status Scale (FSS) of -the Greek- Boston carpal tunnel questionnaire (BCTQ) | 3-7 days after the treatment protocol
  The Boston carpal tunnel questionnaire (BCTQ) is an easy, disease-specific measurement of self-reported symptom severity and functional status for carpal tunnel syndrome (CTS). It has two distinct scales, the Symptom Severity Scale (SSS) which has 11 questions and the Functional Status Scale (FSS) containing 8 questions. Each scale using a five-point rating score generates a final score which ranges from 1 to 5, with the higher indicating greater disability. We will use the Greek version of the BCTQ, which had been examined for reliability and validity and responsiveness before and after the intervention.
change from baseline in Visual Analogue Scale (VAS) | 3-7 days after the treatment protocol
  The Visual Analogue Scale (VAS) will be used to measure the severity of pain induced by carpal tunnel syndrome before and after the intervention. Zero is the minimum score and ten is the maximum score for pain.
change from baseline in median sensory nerve conduction velocity (SNCV) | 3-7 days after the treatment protocol
  Change from baseline of electrophysiological parameters will be assessed after the treatment by using Keypoint electromyography
change from baseline in median distal motor latency (DML) | 3-7 days after the treatment protocol
  Change from baseline of electrophysiological parameters will be assessed after the treatment by using Keypoint electromyography
change from baseline in median sensory nerve action potential (SNAP) | 3-7 days after the treatment protocol
  Change from baseline of electrophysiological parameters will be assessed after the treatment by using Keypoint electromyography
change from baseline in cross sectional area of the median nerve | 3-7 days after the treatment protocol
  The Cross sectional area (CSA) of the median nerve at the inlet of carpal tunnel (at the level of pisiform and scaphoid bone) will be measured before and after treatment by the Sonosite edge Ultrasound machine (6 MHz- 15 MHz linear probe)
adverse events | 3-7 days after the treatment protocol
  number of patients who develop adverse events
number of patients who require medication throughout treatment | 3-7 days after the treatment protocol
  need for additional medication throughout treatment
change from baseline in distal sensory latency (DSL) of the median nerve | 3-7 days after the treatment protocol
  Change from baseline of electrophysiological parameters will be assessed after the treatment by using Keypoint electromyography

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, PhD, DESA, Principal Investigator — Aretaieion University Hospital
Locations (2):
- Greece (2):
  - Pain Clinic of Aretaieion University Hospital, Athens
  - Laboratory of Musculoskeletal Physiotherapy of University of West Attica, Athens

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bougea A, Zambelis T, Voskou P, Katsika PZ, Tzavara C, Kokotis P, Karandreas N. Reliability and Validation of the Greek Version of the Boston Carpal Tunnel Questionnaire. Hand (N Y). 2018 Sep;13(5):593-599. doi: 10.1177/1558944717725379. Epub 2017 Aug 20. PMID 28825339
- [Background] Graham B, Peljovich AE, Afra R, Cho MS, Gray R, Stephenson J, Gurman A, MacDermid J, Mlady G, Patel AT, Rempel D, Rozental TD, Salajegheh MK, Keith MW, Jevsevar DS, Shea KG, Bozic KJ, Adams J, Evans JM, Lubahn J, Ray WZ, Spinner R, Thomson G, Shaffer WO, Cummins DS, Murray JN, Mohiuddin M, Mullen K, Shores P, Woznica A, Linskey E, Martinez Y, Sevarino K. The American Academy of Orthopaedic Surgeons Evidence-Based Clinical Practice Guideline on: Management of Carpal Tunnel Syndrome. J Bone Joint Surg Am. 2016 Oct 19;98(20):1750-1754. doi: 10.2106/JBJS.16.00719. No abstract available. PMID 27869627
- [Background] Jablecki CK, Andary MT, Floeter MK, Miller RG, Quartly CA, Vennix MJ, Wilson JR; American Association of Electrodiagnostic Medicine; American Academy of Neurology; American Academy of Physical Medicine and Rehabilitation. Practice parameter: Electrodiagnostic studies in carpal tunnel syndrome [RETIRED]. Report of the American Association of Electrodiagnostic Medicine, American Academy of Neurology, and the American Academy of Physical Medicine and Rehabilitation. Neurology. 2002 Jun 11;58(11):1589-92. doi: 10.1212/wnl.58.11.1589. No abstract available. PMID 12058083
- [Background] Levine DW, Simmons BP, Koris MJ, Daltroy LH, Hohl GG, Fossel AH, Katz JN. A self-administered questionnaire for the assessment of severity of symptoms and functional status in carpal tunnel syndrome. J Bone Joint Surg Am. 1993 Nov;75(11):1585-92. doi: 10.2106/00004623-199311000-00002. PMID 8245050
- [Background] McCormack HM, Horne DJ, Sheather S. Clinical applications of visual analogue scales: a critical review. Psychol Med. 1988 Nov;18(4):1007-19. doi: 10.1017/s0033291700009934. PMID 3078045
- [Background] Michopoulos I, Douzenis A, Kalkavoura C, Christodoulou C, Michalopoulou P, Kalemi G, Fineti K, Patapis P, Protopapas K, Lykouras L. Hospital Anxiety and Depression Scale (HADS): validation in a Greek general hospital sample. Ann Gen Psychiatry. 2008 Mar 6;7:4. doi: 10.1186/1744-859X-7-4. PMID 18325093
- [Background] Milone MT, Karim A, Klifto CS, Capo JT. Analysis of Expected Costs of Carpal Tunnel Syndrome Treatment Strategies. Hand (N Y). 2019 May;14(3):317-323. doi: 10.1177/1558944717743597. Epub 2017 Nov 22. PMID 29166787
- [Background] Padua L, LoMonaco M, Gregori B, Valente EM, Padua R, Tonali P. Neurophysiological classification and sensitivity in 500 carpal tunnel syndrome hands. Acta Neurol Scand. 1997 Oct;96(4):211-7. doi: 10.1111/j.1600-0404.1997.tb00271.x. PMID 9325471
- [Background] Snaith RP, Zigmond AS. The hospital anxiety and depression scale. Br Med J (Clin Res Ed). 1986 Feb 1;292(6516):344. doi: 10.1136/bmj.292.6516.344. No abstract available. PMID 3080166
- [Background] Wu IX, Lam VC, Ho RS, Cheung WK, Sit RW, Chou LW, Zhang Y, Leung TH, Chung VC. Acupuncture and related interventions for carpal tunnel syndrome: systematic review. Clin Rehabil. 2020 Jan;34(1):34-44. doi: 10.1177/0269215519877511. Epub 2019 Sep 26. PMID 31556315
- [Derived] Ntoutsouli AM, Georgoudis G, Papapostolou A, Karavis M, Petrou DD, Vadalouca A, Theodoraki K. Effects of electroacupuncture on carpal tunnel syndrome: a clinical, electrophysiological and ultrasonographical pilot study. Acupunct Med. 2025 Aug;43(4):198-207. doi: 10.1177/09645284251363989. Epub 2025 Aug 4. PMID 40760926